CLINICAL TRIAL: NCT05510700
Title: Acupuncture for Breast Cancer-related Insomnia : a Multicenter Randomized Controlled Clinical Trial
Brief Title: Efficacy of Acupuncture Treatment for Breast Cancer-associated Insomnia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yin Ping (Other)
Collaborators: Longhua Hospital (Other)
Responsible Party: Sponsor-Investigator, Yin Ping, Shanghai University of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GY202201
Record Dates: First submitted 2022-08-09; First posted 2022-08-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Breast Neoplasms; Insomnia
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture group (Experimental): Participants will be given sleep hygiene instructions. Participants will receive acupuncture treatment at Nei Guan (PC 6), Shen Men (HT 7), Shen Ting (GV 24), Yin Tang (GV 29), Zhong Wan (CV 12), San Yin Jiao (SP 6), Zhao Hai (KI 6), and Shen Mai (BL 62). Among the above acupoints, Nei Guan (PC 6), Shen Men (HT 7), San Yin Jiao (SP 6), Zhao Hai (KI 6), and Shen Mai (BL 62) are all taken from both sides.
  Participants will receive three treatments per week (every other day), each lasting 30 minutes, for a total of 12 sessions over the course of four weeks. The follow-up observation will be recorded on week 8 and 16.
  Interventions: Device: Acupuncture
- Sham acupuncture group (Sham Comparator): Participants will be given sleep hygiene instructions. To match the true acupuncture points, sham treatment at sham Nei Guan (PC 6), Shen Men (HT 7), Shen Ting (GV 24), Yin Tang (GV 29), Zhong Wan (CV 12), San Yin Jiao (SP 6), Zhao Hai (KI 6), and Shen Mai (BL 62) will be used.
  Participants will have the same needle retention time, treatment time, and follow-up time as the acupuncture group.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture — All acupuncture locations will be sterilized on a routine basis. As acupuncture needles are inserted, all points will be lifted, twisted, and stabbed to activate de qi, a sensation generally associated with acupuncture, including swelling, soreness, numbness, and heaviness.
  Arms: Acupuncture group
Device: Sham acupuncture — The placebo needles selected for this study are flat-tipped needles without a tip that cannot be pierced into the skin. Also, an external patch device will hold the needles in place and these needles are visually pierced into the skin. At the end of the treatment, the acupuncturist will press the acupuncture point with a dry cotton ball to allow the patient to feel the "needles" being pulled out.
  Arms: Sham acupuncture group

SUMMARY:
Through a scientific and standardized multicenter, randomized, and controlled study method, the investigators evaluated the clinical efficacy and safety of acupuncture in the treatment of breast cancer-related insomnia, with a view to providing a reliable theoretical basis for the treatment of breast cancer-related insomnia with acupuncture.

DETAILED DESCRIPTION:
Insomnia associated with breast cancer is one of the most common symptoms among breast cancer patients, which seriously affects the life quality of breast cancer patients. Therefore, how to better improve their life quality and insomnia symptoms is of important clinical significance. Previous studies have shown that acupuncture may be beneficial for improving sleep disorders in cancer patients. However, the available clinical evidence is mixed, and clinical studies on acupuncture for breast cancer-associated insomnia lack well-designed, high-quality clinical evidence. The purpose of this study was to evaluate the clinical efficacy and safety of acupuncture for breast cancer-associated insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for breast cancer in the 2022 V2 edition of the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology and the American Joint Committee on Cancer (AJCC) Cancer Staging Manual (8th edition) for breast cancer staging criteria meet the diagnostic criteria for breast cancer with TNM stage I to III; meet the diagnostic criteria for insomnia within the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), and insomnia related to the cancer itself or to cancer-related treatment occurred after breast cancer diagnosis and lasted for at least 1 month.
* Female patients aged 18-75 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Sleep severity index scale (ISI) score ≥ 8.
* Predicted survival of ≥ 6 months.
* Patients had never received acupuncture treatment.
* No mental or intellectual abnormalities, able to understand the provisions of the scales and complete the assessment.
* Consent to participate in this study and sign a written informed consent.

Exclusion Criteria:

* Combination of more serious heart, liver, kidney, and other major diseases. f applicable, indicate if participant eligibility is based on self-representation of gender identity.
* Patients who are pregnant or breastfeeding.
* Those with planned surgery during the trial.
* Previous history of drug abuse or addiction.
* Those who have taken sedative-hypnotic drugs or antipsychotic drugs 2 weeks prior to the baseline visit, or received other treatment for insomnia (e.g., cognitive behavioral therapy, etc.) 3 months prior to the baseline visit, which may affect the efficacy of the observation.
* Insomnia due to cancer pain with an numeric rating scale (NRS) score ≥ 4, or insomnia due to other physical diseases.
* Long-term night work or irregular rest and relaxation.
* Ulcers, abscesses, skin infections, etc. at the site of needling.
* Participation in other clinical medical trial studies within the last month.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment response rate of Insomnia Severity Index (ISI) | Week 4 (end of treatment)
  The percentage of people whose total Insomnia Severity Index (ISI) score decreased by ≥8 points at the end of week 4 treatment compared to the baseline score. The ISI consists of 7 items to assess the nature and symptoms of the subject's sleep disorders. Questions addressed subjects' subjective ratings of sleep quality, including the severity of symptoms, subjects' satisfaction with their sleep patterns, the impact of the degree of insomnia on daily functioning, subjects' awareness of the impact of insomnia on themselves, and their level of frustration due to their sleep disorders. The scores were 0 to 4, with a total score range from 0 to 28. Higher scores indicate more severe insomnia. ISI levels can be classified as no clinically significant insomnia (0 to 7), mild insomnia (8 to 14), moderate insomnia (15 to 21), and severe insomnia (22 to 28).

SECONDARY OUTCOMES:
Treatment remission rate of Insomnia Severity Index (ISI) | Week 4 (end of treatment), week 8 (follow-up), and week 16(follow-up)
  The percentage of people with a total score of <8 points in total Insomnia Severity Index (ISI) score at the end of week 4, 8 and 16 of treatment compared to the baseline score. The ISI consists of 7 items to assess the nature and symptoms of the subject's sleep disorders. Questions addressed subjects' subjective ratings of sleep quality, including the severity of symptoms, subjects' satisfaction with their sleep patterns, the impact of the degree of insomnia on daily functioning, subjects' awareness of the impact of insomnia on themselves, and their level of frustration due to their sleep disorders. The scores were 0 to 4, with a total score range from 0 to 28. Higher scores indicate more severe insomnia. ISI levels can be classified as no clinically significant insomnia (0 to 7), mild insomnia (8 to 14), moderate insomnia (15 to 21), and severe insomnia (22 to 28).
Sleep Efficiency (SE) with Sleep Diary | At baseline, weeks 1, 2, 3, and 4 (end of treatment)
  It will be determined by sleep diary subjectively. Sleep Efficiency(SE) is the percentage of time spent asleep while in bed. It is calculated by (TST / TIB) × 100%. Sleep parameters measured by sleep diary include Sleep Onset Latency (SOL),Wake After Sleep Onset(WASO),Early morning awakening(EMA), and Total Time in Bed (TIB). Total Sleep Time (TST) is calculated by subtracting SOL, WASO and EMA from TIB.
Generalized Anxiety Disorder Scale (GAD-7) | At baseline and week 4 (end of treatment)
  It is a concise anxiety self-assessment instrument consisting of 7 items to assess patients' anxiety over the past two weeks. This questionnaire has a score of 0-3 for each entry and a total score of 21. The scores are 5-9 for mild anxiety, 10-14 for moderate anxiety, and 15-21 for severe anxiety.
Patient Health Questionnaire-9 (PHQ-9) | At baseline and week 4 (end of treatment)
  It is a simple and validated 9-item depression self-assessment tool that assesses patients' depression over the past 2 weeks. Each item is scored 0-3, with a total score of 27. Among them, 5-9 are mild depression, 10-14 are moderate depression, 15-19 are severe depression, and 20-27 are very severe depression.
Quality of Life Core Scale (QLQ-C30) | At baseline and week 4 (end of treatment)
  It contains 30 entries with six dimensions. Widely used in clinical studies, it is currently used to assess the quality of life situation of patients.
Sleep Efficiency (SE) with Actigraphy | At baseline, weeks 1 and 4 (end of treatment)
  The actigraphy device (wGT3X-BT. LLC, Pensacola, USA) can monitor sleep quality objectively. Sleep Efficiency(SE) is the percentage of time spent asleep while in bed. It is calculated by (TST / TIB) × 100%. The actigraphy device record Sleep Onset Latency (SOL),Wake After Sleep Onset(WASO), Early morning awakening(EMA), and Total Time in Bed (TIB). Total Sleep Time (TST) is calculated by subtracting SOL, WASO and EMA from TIB.
Weekly usage of remedial drugs | At weeks 1, 2, 3, and 4 (end of treatment), week 8 (follow-up), and week 16(follow-up)
  The percentage of participants who used emergency drugs.
Incidence of adverse events | During 1-4 weeks
  The adverse events (AEs) assessment aims at evaluating the AEs of acupuncture treatment.
Treatment response rate of Insomnia Severity Index (ISI) at follow-up visits | Week 8 (follow-up), and week 16(follow-up)
  The percentage of people whose total Insomnia Severity Index (ISI) score decreased by ≥8 points at the end of week 8 and 16 of the treatment compared to the baseline score. The ISI consists of 7 items to assess the nature and symptoms of the subject's sleep disorders. Questions addressed subjects' subjective ratings of sleep quality, including the severity of symptoms, subjects' satisfaction with their sleep patterns, the impact of the degree of insomnia on daily functioning, subjects' awareness of the impact of insomnia on themselves, and their level of frustration due to their sleep disorders. The scores were 0 to 4, with a total score range from 0 to 28. Higher scores indicate more severe insomnia. ISI levels can be classified as no clinically significant insomnia (0 to 7), mild insomnia (8 to 14), moderate insomnia (15 to 21), and severe insomnia (22 to 28).
The mean changes of Insomnia Severity Index (ISI) from baseline | Week 4 (end of treatment), week 8 (follow-up), and week 16(follow-up)
  The ISI consists of 7 items to assess the nature and symptoms of the subject's sleep disorders. Questions addressed subjects' subjective ratings of sleep quality, including the severity of symptoms, subjects' satisfaction with their sleep patterns, the impact of the degree of insomnia on daily functioning, subjects' awareness of the impact of insomnia on themselves, and their level of frustration due to their sleep disorders. The scores were 0 to 4, with a total score range from 0 to 28. Higher scores indicate more severe insomnia. ISI levels can be classified as no clinically significant insomnia (0 to 7), mild insomnia (8 to 14), moderate insomnia (15 to 21), and severe insomnia (22 to 28).
Sleep Awakening (SA) with Actigraphy | At baseline, weeks 1 and 4 (end of treatment)
  It is the number of sleep awakenings during the night that recorded with actigraphy device (wGT3X-BT. LLC, Pensacola, USA).
Average Awaken Time (AA) with Actigraphy | At baseline, weeks 1 and 4 (end of treatment)
  It is estimated by (Wake After Sleep Onset(WASO) / Sleep Awakening(SA)) measured in minutes that recorded with actigraphy device (wGT3X-BT. LLC, Pensacola, USA).

CONTACTS AND LOCATIONS:
Overall Officials: YUELAI CHEN, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morin CM, Edinger JD, Beaulieu-Bonneau S, Ivers H, Krystal AD, Guay B, Belanger L, Cartwright A, Simmons B, Lamy M, Busby M. Effectiveness of Sequential Psychological and Medication Therapies for Insomnia Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Nov 1;77(11):1107-1115. doi: 10.1001/jamapsychiatry.2020.1767. PMID 32639561
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Cocks K, King MT, Velikova G, de Castro G Jr, Martyn St-James M, Fayers PM, Brown JM. Evidence-based guidelines for interpreting change scores for the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30. Eur J Cancer. 2012 Jul;48(11):1713-21. doi: 10.1016/j.ejca.2012.02.059. Epub 2012 Mar 12. PMID 22418017
- [Background] Meltzer LJ, Montgomery-Downs HE, Insana SP, Walsh CM. Use of actigraphy for assessment in pediatric sleep research. Sleep Med Rev. 2012 Oct;16(5):463-75. doi: 10.1016/j.smrv.2011.10.002. Epub 2012 Mar 15. PMID 22424706
- [Derived] Yin P, Fan Q, Liu L, Yang M, Zhang S, Li X, Hou W, Feng Q, Wang X, Jin Z, Li F, Chen Y. Efficacy of acupuncture treatment for breast cancer-related insomnia: study protocol for a multicenter randomized controlled trial. Front Psychiatry. 2024 May 23;15:1301338. doi: 10.3389/fpsyt.2024.1301338. eCollection 2024. PMID 38846918